CLINICAL TRIAL: NCT05864599
Title: External Validation of Uromonitor as a Biomarker for Optimization of NMIBC Management by the CUETO Group
Acronym: EVALUATION
Status: Active, not recruiting | Type: Observational
Sponsor: Pharmalink (Industry)
Responsible Party: Sponsor
Other Study IDs: PIEM-AEU-2023-0001
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Independent validation of Uromonitor as a non-invasive biomarker of recurrence of Non Muscle Invasive Bladder Cancer

DETAILED DESCRIPTION:
This study is intended as an independent validation series for previous studies performed in several European centers with less statistical power. We expect to validate the results from a previous study, reaching the sensitivity and specificity data obtained at generation and first external validation papers. The overall goal of this study is to perform a bigger external multicenter validation study to evaluate the sensitivity, specificity, NPV and PPV of Uromonitor for the detection of bladder cancer recurrence in an independent series of patients.

The specific objectives of this study protocol are the following:

Main endpoint:

• To evaluate the clinical sensitivity, specificity, NPV and PPV of Uromonitor in the detection of bladder cancer recurrence in patients previously diagnosed (over the last 3 months to 2 years) of NMIBC, treated or not, by testing a total of 600 patients (EVALUATION-CUETO Study)

ELIGIBILITY:
Inclusion Criteria:

Main Outcome:

* Age >22.
* Patients with a history of non-muscle invasive bladder cancer (any risk group, any intravesical adjuvant treatment received) over the last 3 months to 2 years, initial or recurrent, undergoing regular cystoscopic surveillance. The criteria for cystoscope FU schedule has been already described in Methods following EAU 2022 Guidelines´ recommendations and related to initial NMIBC risk grouping.
* Patient must be able to provide at least 10 ml of urine.
* Additional 10 ml of urine needs to be collected for cytology.
* Patients must be able to provide informed consent

  2.- Subgroup analysis (secondary Objective 1):
* Age >22
* Patients with a history of primary non-muscle invasive bladder cancer with presence of CIS over the last 3 months to 3 years, and previously treated with BCG undergoing regular cystoscopic surveillance.
* Patient must be able to provide at least 10 ml of urine.
* Additional 10 ml of urine needs to be collected for cytology.
* Patients must be able to provide informed consent.

  3.- Subgroup analysis (secondary Objective 2):
* Age >22
* Patients included in both previous groups, having a positive Uromonitor® test and a negative cystoscopy to be followed by two years as previously described depending on initial NMIBC risk group. The rest of the patients will also be followed 2 years to detect later recurrences/progression figures.

Exclusion Criteria:

* Patients who are unable to provide the minimum amount of urine needed to perform one test.

  * Patients planning to undergo radical cystectomy or chemotherapy, radiation for UC
  * Patients at risk for non-definitive information derived from the cystoscope due to different conditions:
* Not possible to ascertain informative cystoscope due to intolerance to the procedure
* Presence of bladder stone
* Presence of entero-vesical fistulae
* Presence of vesico-vaginal fistulae
* Non informative cystoscope due to macroscopic haematuria or cloudy urine
* Other conditions avoiding a clear tumour rule-out cystoscope

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of non-muscle invasive bladder cancer (any risk group, any intravesical adjuvant treatment received) over the last 3 months to 2 years, initial or recurrent, undergoing regular cystoscopic surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, NPV and PPV of Uromonitor | 2 years after diagnosis
  To evaluate the clinical sensitivity, specificity, NPV and PPV of Uromonitor in the detection of bladder cancer recurrence in patients previously diagnosed (over the last 3 months to 2 years) of NMIBC, treated or not

SECONDARY OUTCOMES:
Statistics in CIS, treated or not | 2 years after diagnosis
  To evaluate the clinical sensitivity and specificity of Uromonitor in the detection of bladder cancer recurrence in patients previously diagnosed (over the last 3 months to 3 years) of NMIBC with carcinoma in situ (CIS) associated and treated with BCG
Early diagnostics | 4 years after diagnosis
  To check if Uromonitor can provide some early diagnostics of NIMBC by following for two years a group of false positive patients of both previous groups (Uromonitor Positive / Cystoscopy Negative)

CONTACTS AND LOCATIONS:
Overall Officials: José Rubio-Briones, MD PhD, Principal Investigator — Hospital 9 d'Octubre
Locations (1):
- Hospital Vithas 9 d'Octubre, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided